CLINICAL TRIAL: NCT05015946
Title: Handball-based Exercise for People Diagnosed With Type 2 Diabetes: a Feasibility Study
Brief Title: Handball-based Exercise and Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College of Northern Denmark (Other)
Collaborators: Danish Handball Federation (Unknown); The Danish Diabetes Association (Other); Research Unit for General Practice in Aalborg (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCN-FoU-24000473
Record Dates: First submitted 2021-06-03; First posted 2021-08-23 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2020-09

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes Mellitus; Glucose Metabolism Disorder; Metabolic Diseases; Endocrine System Disease; Team Handball Training; Team Sport
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases

STUDY DESIGN:
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Small-sided team handball training (Experimental): 60 minutes small-sided team handball training. Initial 20 minutes of warm-up including exercises for strength, aerobic, balance, coordination, and mobility. Hereafter 20 minutes of handball specific exercises including dribbling, running and shooting. Final 20 minutes of small-sided handball matches.
  Interventions: Behavioral: Small-sided team handball training

INTERVENTIONS:
Behavioral: Small-sided team handball training — 60 minutes small-sided team handball training. Initial 20 minutes of warm-up including exercises for strength, aerobic, balance, coordination, and mobility. Hereafter 20 minutes of handball specific exercises including dribbling, running and shooting. Final 20 minutes of small-sided handball matches.

SUMMARY:
This single-arm pilot study aims to investigate the feasibility of a handball-based intervention to people diagnosed with type 2 diabetes, including monitoring aerobic intensities and movement strategies during the intervention, and monitoring recruitment, adherence, and adverse events.

Furthermore, the study aims to investigate the feasibility of a test battery including both physiological and patient-reported outcomes, and to investigate preliminary exercise effects.

DETAILED DESCRIPTION:
Physical activity and exercise are known to be beneficial for increasing insulin sensitivity in skeletal muscle in healthy as well as in individuals with type 2 diabetes. But many patients who recently have been diagnosed with type-2 diabetes is often living a sedentary lifestyle and have poor adherence to physical interventions.

High intensity interval training as well as team-based interventions has proven to be effectful in regulation of physiological parameters related to type 2 diabetes. The aim of this study is to investigate the feasibility of a handball-based intervention to people diagnosed with type 2 diabetes

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes
* Understands and speaks danish

Exclusion Criteria:

* If General Practitioner do not recommend participation in the intervention

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
Concentration of Hemoglobin A1c (HbA1c) (mmol/mol) | change from baseline to 12 weeks
  HbA1c measured with HemoCue HbA1c 501
Peak oxygen uptake (VO2peak) | change from baseline to 12 weeks
  Peak oxygen uptake measured with incremental cycling test
Health related quality of life (HRQoL) | change from baseline to 12 weeks
  Health related quality of life measured with the danish version of Short Form 36 (SF-36)

SECONDARY OUTCOMES:
Concentration of Cholesterol | change from baseline to 12 weeks
  Total cholesterol, low density lipoprotein (LDL), high density lipoprotein (HDL) measured with Accutrend Plus Cholesterol Meter
Body mass index (BMI) | change from baseline to 12 weeks
  Body mass index measured by kg/M2
Body fat mass (kg) | change from baseline to 12 weeks
  Total body fat in kg measured with Tanita MC-180MA, Tokyo, Japan
Lean body mass (kg) | change from baseline to 12 weeks
  Lean body mass in kg measured with Tanita MC-180MA, Tokyo, Japan
Visceral fat (hip/waist ratio) | change from baseline to 12 weeks
  Visceral adipose tissue measured with hip (widest part of the hip) and waist (2.5 cm above the navel) ratio.
Blood pressure and resting puls | change from baseline to 12 weeks
  Blood pressure and resting puls measured with an automatic upperarm blood pressure monitor
Aerobic performance test (aerobic endurance) | change from baseline to 12 weeks
  Aerobic endurance measured with Intermittent Recovery Test Level 1
Self-care behavior | change from baseline to 12 weeks
  Self-care behavior measured with diabetes Intention, Attitude, and Behavior Questionnaire (DIAB-Q)
Physical activity levels | change from baseline to 12 weeks
  Physical activity scale (PAS)
Aerobic intensity and movement patterns | measured during intervention in week 2,3,6,7,10 and 11.
  Aerobic intensities (percent of maximal heart rate) measured with pulse monitor, and movement patterns (Metabolic Equivalent of Task (MET)) measured with accelerometer.

CONTACTS AND LOCATIONS:
Locations (1):
- The Department of Physiotherapy, University College of Northern Denmark, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No